CLINICAL TRIAL: NCT01662908
Title: A Randomized, Open-Label, Parallel-Group, Multi-Center Study for the Evaluation of Efficacy and Safety of Edoxaban Monotherapy Versus (LMW) Heparin/Warfarin in Subjects With Symptomatic Deep-Vein Thrombosis - Edoxaban Thrombus Reduction Imaging Study
Brief Title: A Randomized, Open-Label, Parallel-Group, Multi-Center Study for the Evaluation of Efficacy and Safety of Edoxaban Monotherapy Versus Low Molecular Weight (LMW) Heparin/Warfarin in Subjects With Symptomatic Deep-Vein Thrombosis
Acronym: eTRIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DU176b-D-U211
Record Dates: First submitted 2012-08-02; First posted 2012-08-13 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2017-05

CONDITIONS: Deep Vein Thrombosis; Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — edoxaban; Enoxaparin; Heparin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- edoxaban tosylate (Experimental)
  Interventions: Drug: edoxaban tosylate
- heparin/warfarin (Active Comparator)
  Interventions: Drug: enoxaparin/unfractionated heparin; Drug: warfarin

INTERVENTIONS:
Drug: edoxaban tosylate — edoxaban tosylate (DU-176b), film-coated for oral use, 90 mg once daily (QD) for 10 days (±2 days) followed by 60 mg QD for a total of approximately 90 days of edoxaban treatment
  Arms: edoxaban tosylate
Drug: enoxaparin/unfractionated heparin — enoxaparin - administered by subcutaneous injection;1 mg/kg/ twice daily or 1.5 mg/kg once daily unfractionated heparin - started with 5000 IU bolus intravenous administration, 1300 IU/h continuous infusion, minimum of 5 days of treatment and stopped when target INR (2.0 - 3.0) is achieved.
  Arms: heparin/warfarin
Drug: warfarin — tablet for oral use; daily dosage, adjusted to maintain international normalized ratio (INR) between 2.0 and 3.0; 90 days treatment.
  Arms: heparin/warfarin

SUMMARY:
Assess the relative change in thrombus volume as determined by two assessments (Baseline and Day 14-21) with magnetic resonance venography (MRV) in subjects with deep-vein thrombosis (DVT) treated with either an edoxaban monotherapy regimen or a low molecular weight (LMW) heparin/warfarin regimen.

DETAILED DESCRIPTION:
The classical management of patients with venous thromboembolism (VTE) consists of an initial treatment of at least five days of a (LMW) heparin followed by long-term treatment with a vitamin K antagonist (VKA), such as warfarin. The eTRIS study will address the clinically important question of whether edoxaban monotherapy, without concomitant (LMW) heparin at the time of treatment initiation is comparable to or better than standard treatment with (LMW) heparin/warfarin therapy in subjects with acute symptomatic DVT as assessed by the relative change from baseline in thrombus volume (measured by MRI) at Day 14-21.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects older than the minimum legal adult age (country specific)
* Acute symptomatic proximal DVT involving the popliteal, femoral or iliac veins confirmed by compression ultrasonography (CUS) or other appropriate imaging techniques (such as venography or spiral/contrast CT) with symptom onset < or = 1week prior to randomization
* Able to provide signed informed consent

Exclusion Criteria:

* Concomitant pulmonary embolism known to the investigator at the time of randomization
* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of DVT
* Indication for warfarin other than DVT
* More than 48 hours pre-treatment with therapeutic dosages of anti-coagulant treatment [low molecular weight heparin (LMWH), unfractionated heparin (UFH), fondaparinux, VKA, factor Xa inhibitor or other anti coagulant per local labeling] prior to randomization to treat the current episode
* Treatment with any investigational drug within 30 days prior to randomization
* Calculated creatinine clearance (CrCL) < 30 mL/min
* Significant liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis) or alanine aminotransferase (ALT) > or = 2 times the upper limit of normal (ULN), or total bilirubin (TBL) > or = to 1.5 times the ULN (however subjects whose elevated TBL is due to known Gilbert's syndrome may be included in the study)
* Subjects with active cancer for whom long term treatment with (LMW) heparin is anticipated
* Life expectancy < 3 months
* Active bleeding or high risk for bleeding contraindicating treatment with (LMW) heparin or warfarin
* Uncontrolled hypertension as judged by the Investigator (e.g., systolic blood pressure > 170 mmHg or diastolic blood pressure > 100 mmHg despite antihypertensive medications confirmed by repeat measurement)
* Women of childbearing potential without proper contraceptive measures (i.e., a method of contraception with a failure rate < 1 % during the course of the study including the observational period) and women who are pregnant or breast feeding
* Any contraindication listed in the local labeling of LMWH, UFH, or warfarin
* Chronic treatment with non-aspirin non-steroidal anti-inflammatory drugs (NSAIDs) including both cyclooxygenase-1 (COX-1) and cyclooxygenase-2 (COX- 2) inhibitors for > or = 4 days/week anticipated to continue during the study.
* Treatment with aspirin in a dosage of more than 100 mg/per day or dual antiplatelet therapy (any two antiplatelet agents including aspirin plus any other oral or intravenous [IV] antiplatelet drug) anticipated to continue during the study
* Treatment with P-gp inhibitors is not permitted at the time of randomization; subsequent use is permitted, with a dose reduction in the edoxaban monotherapy treatment arm.
* Known history of positive Hepatitis B antigen or Hepatitis C antibody
* Subjects with any condition that, as judged by the investigator, would put the subject at increased risk of harm if he/she participated in the study; including, but not limited to, subjects at increased risk of harm if given a gadolinium-based contrast agent such as gadofosveset trisodium (Ablavar®)
* Subjects for whom MRI would be contraindicated (e.g., subjects with metal implants) or for whom the use of a gadolinium-based contrast agent such as gadofosveset trisodium (Ablavar®) would be contraindicated
* Subject has previously entered this study or another edoxaban study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (34):
- United States (29):
  - Dothan, Alabama
  - Montgomery, Alabama
  - Sacramento, California
  - Atlantis, Florida
  - Clearwater, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Jonesboro, Georgia
  - Lafayette, Indiana
  - Paducah, Kentucky
  - Covington, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Randallstown, Maryland
  - Butte, Montana
  - Grand Island, Nebraska
  - Rochester, New York
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Wilmington, North Carolina
  - Maumee, Ohio
  - Camp Hill, Pennsylvania
  - Ephrata, Pennsylvania
  - Sellersville, Pennsylvania
  - Rapid City, South Dakota
  - Fredericksburg, Virginia
  - Tacoma, Washington
- Canada (5):
  - Edmonton, Alberta
  - London, Ontario
  - Newmarket, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Piazza G, Mani V, Goldhaber SZ, Grosso MA, Mercuri M, Lanz HJ, Schussler S, Hsu C, Chinigo A, Ritchie B, Nadar V, Cannon K, Pullman J, Concha M, Schul M, Fayad ZA; edoxaban Thrombus Reduction Imaging Study (eTRIS) Investigators. Magnetic resonance venography to assess thrombus resolution with edoxaban monotherapy versus parenteral anticoagulation/warfarin for symptomatic deep vein thrombosis: A multicenter feasibility study. Vasc Med. 2016 Aug;21(4):361-8. doi: 10.1177/1358863X16645853. Epub 2016 May 10. PMID 27165711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2012 through January 2014, a total of 85 patients were enrolled at 26 centers in North America (US and Canada). One subject was not included in either the full analysis set or the safety analysis set because of major protocol violation - he did not take any dose of study drug.
Groups:
- Edoxaban: Participants treated with edoxaban
- Warfarin: Participants treated with warfarin
Period: Overall Study
Arm/Group | Edoxaban | Warfarin
Started | 56 | 28
Completed | 50 | 23
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edoxaban | Warfarin | Total
Number analyzed (Participants) | 56 | 28 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 22 | 63
  >=65 years | 15 | 6 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 41 | 21 | 62
Region of Enrollment [Number; unit: participants]
  Canada | 16 | 6 | 22
  United States | 40 | 22 | 62

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Thrombus Volume Assessed by MRI [Using the Magnetic Resonance Venography (MRV) Method]
Description: Thrombus Volume (mm^3) was measured at baseline and between days 14 to 21 using MRI results as determined by Magnetic Resonance Venography (MRV) method, and the relative percentage change from baseline was calculated
Time Frame: Baseline to final visit (Day 14-21)
Population: Modified intention to treat (mITT), defined as intention to treat minus the one patient who did not take the investigational product
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Edoxaban | Warfarin
Number analyzed (Participants) | 56 | 28
percentage of change | -46.6 (45.53) | -51.4 (32.96)
Statistical Analysis 1: Comparison: Edoxaban vs Warfarin; Test type: Other; Mean Difference (Final Values) = 8.8, 95% CI 2-sided [-12.7 to 30.2], Standard Error of Mean 10.74

2. Secondary Outcome: Number of Participants With Clinically Relevant Bleeding
Description: Clinically relevant bleeding was defined as major or clinically relevant non-major bleeding
Time Frame: Initial dose of study drug up to 3 days after last dose
Population: Adjudicated in the mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Warfarin
Number analyzed (Participants) | 56 | 28
Participants | 3 | 2

3. Secondary Outcome: Number of Participants With Recurrence of Venous Thromboembolism (VTE)
Description: Number of participants with investigator-confirmed recurrent VTE events that start or worsen after the first dose of study drug and prior to the date of the final visit or telephone contact (inclusive)
Time Frame: Baseline to final visit (Day 14-21)
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Warfarin
Number analyzed (Participants) | 56 | 28
Participants | 4 | 2

4. Secondary Outcome: Number of Participants With Major Adverse Cardiovascular Events (MACE)
Description: MACE is defined as a composite of non-fatal myocardial infarction (MI), non-fatal stroke, non-fatal systemic embolic event (SEE) and cardiovascular death
Time Frame: Initial dose of study drug up to 3 days after last dose
Population: Adjudicated confirmed events in the mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Warfarin
Number analyzed (Participants) | 56 | 28
Participants | 2 | 0

5. Secondary Outcome: Number of Participants With Change From Baseline in the Presence or Absence of Thrombus by Vessel
Time Frame: Baseline to final visit (Day 14-21)
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Warfarin
Number analyzed (Participants) | 56 | 28
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Edoxaban | Warfarin
Serious Adverse Events (participants affected / at risk) | 4/56 | 4/28
Other Adverse Events (participants affected / at risk) | 32/56 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban (N=56) | Warfarin (N=28)
Bronchitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban (N=56) | Warfarin (N=28)
Urinary Tract Infection (Infections and infestations) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Neuritis (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Skln ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Renal cyst (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 2
Fatigue (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 0
Injection site haematoma (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Epstein-Barr virus antibody positive (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1
Arthopod bite (Injury, poisoning and procedural complications) | 1 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other